CLINICAL TRIAL: NCT00582049
Title: Research on the Environment and Children's Health: Retinoblastoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Pennsylvania (Other); New York Presbyterian Hospital (Other); Milton S. Hershey Medical Center (Other)
Responsible Party: Ira Dunkel, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 03-030
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma; Sporadic heritable retinoblastoma; Paternal exposures
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (2):
- 1: Cases: retinoblastoma patients
- 2: Controls: first cousins or other blood relatives of the retinoblastoma patients (relative controls) or friends of the retinoblastoma patients or children of friends of the parents (friend controls).

SUMMARY:
The purpose of the research study is to learn more about the causes of retinoblastoma and to identify possible risk factors in the parents of patients with retinoblastoma. This kind of study is called an epidemiology study and is often done by interviewing people with and without the disease. In the case of a childhood disease, the researchers ask about experiences of the parents and children before the disease developed.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the role of paternal exposures in the etiology of sporadic heritable retinoblastoma (RBL). The study has a matched case-control design with a sample size of 255 pairs. Cases will be children with sporadic heritable (RBL) identified from eight hospitals that together treat most of the RBL patients in the U.S. and Canada. We will use regional controls matched on year of birth and state/province of residence identified by randomdigit-dialing (RDD). Fathers and mothers of cases and controls will be interviewed by telephone about their occupational, medical, dietary, and personal exposures before the index child's conception. Blood samples will be obtained on cases and their parents for DNA isolation. The case's DNA will be used to characterize the disease-causing RB1 mutation. The parent's DNA will be used to detect the few instances in which a parent also has the RB1 mutation, i.e., the child's RBL is familial rather than sporadic.

ELIGIBILITY:
Inclusion Criteria:

* Cases will be children with sporadic heritable RBL, i.e., bilateral RBL without a family history of the disorder.
* Cases will be diagnosed with retinoblastoma in an approximately 7-year period, beginning January 1, 1998 and continuing until the sample size is reached.
* The case family must reside in the continental U.S., Alaska, or Canada.
* The case family must have a telephone in the household.
* The patient's physician must give permission to contact the parents of the case.
* The biologic father or mother of the case must be available and consent to be interviewed.
* The father or mother must speak English or Spanish.
* Genetic counseling regarding RB1 gene mutation analysis must be done prior to registration onto study.

Exclusion Criteria:

- Cases that do not meet the above criteria will be ineligible to participate and excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects (cases) will be children with sporadic heritable RBL and their parents. Parents of children without RBL will be identified and will participate as controls.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2003-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
demographic and exposure information by telephone interview | 5 years 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org